CLINICAL TRIAL: NCT00946231
Title: HF Assessment With BNP In The Home
Brief Title: Heart Failure (HF) Assessment With B-type Natriuretic Peptide (BNP) In The Home
Acronym: HABIT
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Collaborators: Inverness Medical Innovations (Industry)
Responsible Party: Clinical Study Manager, Biosite Incorporated
Other Study IDs: BSTE-0108
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; BNP; B-type natriuretic peptide; home testing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Subjects admitted to the hospital with decompensated heart failure.

SUMMARY:
The HABIT clinical study is being performed to determine the benefit and optimal frequency for at home testing of B-type natriuretic peptide (BNP) for heart failure patients following hospitalization from decompensation. Subjects will be enrolled following hospitalization for decompensated heart failure. Enrolled subjects will be trained on the use of the Triage Touch meter for fingerstick BNP assessment; these subjects will then test their BNP levels daily using the Triage Touch product for approximately 60 days.

DETAILED DESCRIPTION:
This is a multi-center, single-arm double-blinded prospective clinical study to determine the optimal frequency of home B-type natriuretic peptide (BNP) testing and the changes in BNP concentrations that correlate with clinical heart failure (HF) decompensation and related adverse clinical outcomes in at-risk HF patients. Approximately 200 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older);
* Admitted to the hospital or observation unit with a diagnosis of decompensated HF for which treatment will be administered;
* Blood BNP level measurement > 400 pg/mL documented during admission; If NT-proBNP is used routinely in the laboratory at a clinical site rather than BNP, then blood NT-proBNP level measurement > 1,600 pg/mL documented during admission.
* Successfully trained on how to perform a fingerstick and to use the Triage touch.
* Either the subject or their care provider is fluent in reading and writing English

Exclusion Criteria:

* Unwilling or unable to provide written informed consent;
* Acute coronary syndrome (ACS) that is concomitant with the diagnosis of decompensated HF and for which treatment will be provided.

A history of ACS is not reason for exclusion if it is not concomitant with the present decompensated HF for which admission is being made. Small elevations in cardiac troponin that are considered by the treating physician to be associated with myocardial injury due to the acute decompensated HF and not due to a concomitant ACS or myocardial infarction are not a basis for exclusion.

* Previous cardiac transplantation - or cardiac transplantation anticipated within 3 months;
* Current or planned use of a left ventricular assist device (LVAD), use of outpatient intravenous inotropic HF therapy, major surgical procedure or percutaneous coronary intervention within 3 months;
* Life expectancy less than 3 months due to causes other than HF or cardiovascular disease (e.g., cancer);
* End stage renal disease;
* Prisoner or other institutionalized or vulnerable individual;
* Residence in regions where either transmission of Triage Touch data or a home visit on day 5 is not possible.
* Dementia, tremors or other impediments to performing daily home BNP testing via fingerstick.
* Deemed by the Investigator not to be likely to comply with study-mandated procedures or instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted to the hospital with decompensated Heart Failure. Subjects may be enrolled while still in the hospital or within 3 days post-discharge through a heart failure clinic or other type of outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To use the Triage touch to determine the optimal frequency of home BNP testing and the changes in BNP concentrations that correlate with clinical HF decompensations and related adverse events in at-risk HF patients. | Day 5, Day 30 and Day 60

SECONDARY OUTCOMES:
To determine the feasibility of frequent home BNP self-testing with the Triage touch in the study population. | Day 5, Day 30 and Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Maisel, MD, Principal Investigator — Veterans Affairs San Diego Healthcare System
Locations (11):
- United States (11):
  - Care Clinical Research Corp DBA Beaver Medical Center, Banning, California
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda VA Medical Center, Loma Linda, California
  - Mission Internal Medical Group, Mission Viejo, California
  - St. Josephs Hospital, Orange, California
  - University of California Irvine Medical Center, Orange, California
  - Desert Cardiology Center, Rancho Mirage, California
  - UCSD Medical Center, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - VA- UCSD, San Diego, California

REFERENCES:
- [Derived] Maisel A, Barnard D, Jaski B, Frivold G, Marais J, Azer M, Miyamoto MI, Lombardo D, Kelsay D, Borden K, Iqbal N, Taub PR, Kupfer K, Clopton P, Greenberg B. Primary results of the HABIT Trial (heart failure assessment with BNP in the home). J Am Coll Cardiol. 2013 Apr 23;61(16):1726-35. doi: 10.1016/j.jacc.2013.01.052. Epub 2013 Mar 26. PMID 23500322